CLINICAL TRIAL: NCT01148797
Title: A 6 Month Phase 2, Multi-Center, Open-label, Single Arm Study to Evaluate the Safety and Efficacy of Treatment With Canakinumab in Pediatric Patients With Colchicine Intolerant or Colchicine Resistant Familial Mediterranean Fever
Brief Title: Evaluate the Safety and Efficacy of Canakinumab in Pediatric Patients With Colchicine Intolerant or Colchicine Resistant Familial Mediterranean Fever (FMF)
Acronym: CONTROL FMF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACZ885D2204
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Colchicine Resistant/Intolerant Familial Mediterranean Fever
Keywords: FMF, Colchicine resistant; Colchicine intolerant; Flare rate; Canakinumab
MeSH Terms: interventions — canakinumab

ARMS (1):
- Canakinumab (Experimental)
  Interventions: Drug: Canakinumab

INTERVENTIONS:
Drug: Canakinumab

SUMMARY:
A study designed to evaluate the role of treatment with a biological agent - Canakinumab in pediatric (age 4-20) Familial Mediterranean Fever (FMF) patients that are intolerant or resistant for colchicine treatment.

The study hypothesis is that Canakinumab will reduce attack frequency and severity.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between 4 and 20 years of age with active type 1 FMF disease (according to Tel-Hashomer Long criteria for diagnosis of FMF) and genetic confirmation of diagnosis (for the study - genetic confirmation is defined as either homozygous or compound heterozygous).
2. Subjects must have type 1 disease characterized by recurrent and short episodes of inflammation and serositis, with an average of at least 3 well documented acute FMF attacks during the previous 3 months that are confirmed by the treating physician, lasting less then a week, and a minimum 14 day- attack free interval between attacks.
3. Subjects must have received an adequate trial of colchicine, defined as treatment of at least 1-2 mg/d (based on subjects age) for at least 3 months, or an inability to tolerate colchicine due to adverse effects in a dose that controls acute attacks in the frequency of less than one attack per month.
4. Subjects treated with anti-IL-1 therapies must complete washout and have experienced at least 2 attacks since (e.g. Anakinra: 3 day washout; Rilonacept: 4 week washout)
5. Subjects treated with anti-TNF drugs must undergo appropriate washout. Prior to randomization, use of Etanercept must be discontinued for 4 weeks or use of Adalimumab or Infliximab must be discontinued for 8 weeks - a full list of washout periods for current treatments will be supplied
6. If subject is a female of childbearing potential, she must agree to use adequate contraception (adequate contraception can include abstinence) for the duration of the trial and 3 months after, and must have a negative serum or urine pregnancy test prior to administration of each dose of study medication.
7. Subject's parent or legal guardian has provided written informed consent prior to screening for this study, or if subject is older than 18 years has provided informed consent him/herself.

Exclusion Criteria:

1. Patients with end-organ dysfunction due to amyloidosis (e.g. existing biopsy proven amyloidosis or proteinuria > 0.5 gram per day)
2. Subjects taking oral or IV steroids within 1 month prior to baseline. Subjects taking steroids for reasons other than FMF - may be enrolled into the study based on discussion with the investigator and sponsor.
3. Presence or history of any other inflammatory rheumatic disease
4. The subject has active non-infective GI disease (e.g., inflammatory bowel disease), a chronic or acute renal or hepatic disorder, or a significant coagulation defect.
5. The subject has an AST (SGOT), ALT (SGPT) or BUN >2 x ULN or creatinine >1.5 mg/dL, and any other laboratory abnormality considered by the examining physician to be clinically significant within 28 days before the Baseline visit.
6. Positive PPD test (according to local guidance) where a latent or active TB infection cannot be excluded via QuantiFERON (T-Spot or radiographic imaging if needed) or via Chest x-ray.
7. The subject has positive human immunodeficiency virus (HIV) status or current (acute or chronic) hepatitis B or C
8. Subjects who are pregnant or lactating
9. Presence of any active or chronic infection or any major episode of infection requiring hospitalization or treatment with i.v. antibiotics within 30 days or oral antibiotics within 14 days prior to screening
10. Malignancy, except for successfully excised squamous or basal cell carcinoma of the skin
11. The subject has received any investigational medication within 30 days before the first dose of study medication or is scheduled to receive an investigational drug, other than study medications described in this protocol, during the course of the study.
12. The subject has received a live virus vaccine within 3 months prior to the baseline visit.
13. Any concurrent medical condition which would, in the investigator's opinion, compromise the subject's ability to tolerate the study drug or would make the subject unable to follow with the protocol.
14. History of/or current psychiatric illness that would interfere with ability to comply with protocol requirements or provide informed consent.
15. Subject has a history of alcohol or drug abuse within the past 6 months that would interfere with ability to comply with protocol requirements.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
To measure the effect of canakinumab on the frequency of FMF attacks, defined as percentage of subjects with at least 50% reduction in the attack frequency during a 3 month treatment period | 0-3 months

SECONDARY OUTCOMES:
To assess the effect of canakinumab with regard to percentage of subjects with no attacks during the 3 months treatment period | 0-3 months
To evaluate the safety and tolerability of canakinumab by monitoring adverse events (AEs) and subject discontinuations due to an AE | 3 months
To assess the change in frequency of FMF attacks during the treatment period | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Eliad Ben Dayan, Study Chair — Novartis Pharmaceuticals
Locations (5):
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center Kfar Saba, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - The Chaim Sheba Medical Center, Ramat Gan

REFERENCES:
- [Background] Lidar M, Livneh A. Familial Mediterranean fever: clinical, molecular and management advancements. Neth J Med. 2007 Oct;65(9):318-24. PMID 17954950
- [Background] Bhat A, Naguwa SM, Gershwin ME. Genetics and new treatment modalities for familial Mediterranean fever. Ann N Y Acad Sci. 2007 Sep;1110:201-8. doi: 10.1196/annals.1423.022. PMID 17911435
- [Background] Mor A, Shinar Y, Zaks N, Langevitz P, Chetrit A, Shtrasburg S, Rabinovitz E, Livneh A. Evaluation of disease severity in familial Mediterranean fever. Semin Arthritis Rheum. 2005 Aug;35(1):57-64. doi: 10.1016/j.semarthrit.2005.02.002. PMID 16084225
- [Background] Masters SL, Simon A, Aksentijevich I, Kastner DL. Horror autoinflammaticus: the molecular pathophysiology of autoinflammatory disease (*). Annu Rev Immunol. 2009;27:621-68. doi: 10.1146/annurev.immunol.25.022106.141627. PMID 19302049
- [Background] Soylemezoglu O, Arga M, Fidan K, Gonen S, Emeksiz HC, Hasanoglu E, Buyan N. Unresponsiveness to colchicine therapy in patients with familial Mediterranean fever homozygous for the M694V mutation. J Rheumatol. 2010 Jan;37(1):182-9. doi: 10.3899/jrheum.090273. Epub 2009 Dec 15. PMID 20008920
- [Background] Roldan R, Ruiz AM, Miranda MD, Collantes E. Anakinra: new therapeutic approach in children with Familial Mediterranean Fever resistant to colchicine. Joint Bone Spine. 2008 Jul;75(4):504-5. doi: 10.1016/j.jbspin.2008.04.001. Epub 2008 Jun 9. PMID 18541452
- [Background] Kuijk LM, Govers AM, Frenkel J, Hofhuis WJ. Effective treatment of a colchicine-resistant familial Mediterranean fever patient with anakinra. Ann Rheum Dis. 2007 Nov;66(11):1545-6. doi: 10.1136/ard.2007.071498. No abstract available. PMID 17934085
- [Background] Moser C, Pohl G, Haslinger I, Knapp S, Rowczenio D, Russel T, Lachmann HJ, Lang U, Kovarik J. Successful treatment of familial Mediterranean fever with Anakinra and outcome after renal transplantation. Nephrol Dial Transplant. 2009 Feb;24(2):676-8. doi: 10.1093/ndt/gfn646. Epub 2008 Nov 25. PMID 19033248
- [Background] Lachmann HJ, Kone-Paut I, Kuemmerle-Deschner JB, Leslie KS, Hachulla E, Quartier P, Gitton X, Widmer A, Patel N, Hawkins PN; Canakinumab in CAPS Study Group. Use of canakinumab in the cryopyrin-associated periodic syndrome. N Engl J Med. 2009 Jun 4;360(23):2416-25. doi: 10.1056/NEJMoa0810787. PMID 19494217
- [Background] Manuel O, Kumar D. QuantiFERON-TB Gold assay for the diagnosis of latent tuberculosis infection. Expert Rev Mol Diagn. 2008 May;8(3):247-56. doi: 10.1586/14737159.8.3.247. PMID 18598104
- [Result] Brik R, Butbul-Aviel Y, Lubin S, Ben Dayan E, Rachmilewitz-Minei T, Tseng L, Hashkes PJ. Canakinumab for the treatment of children with colchicine-resistant familial Mediterranean fever: a 6-month open-label, single-arm pilot study. Arthritis Rheumatol. 2014 Nov;66(11):3241-3. doi: 10.1002/art.38777. No abstract available. PMID 25049046